CLINICAL TRIAL: NCT04169659
Title: Kyphoplasty With Structured Titanium Spheres: Pilot Study. P.R.O.B.E. Trial (Prospective Randomized Open Blinded End Point)
Brief Title: Kyphoplasty With Structured Titanium Spheres
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ARNAS Civico Di Cristina Benfratelli Hospital (Other)
Responsible Party: Principal Investigator, Gabriele Costantino, Principal Investigator, ARNAS Civico Di Cristina Benfratelli Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 232 Civico 2018; MTOrtho (Other: MTOrtho)
Record Dates: First submitted 2019-07-06; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Vertebral Fracture
Keywords: Kyphoplasty; EBM; Titanium; Microsphere; Vertebral fracture
MeSH Terms: conditions — Spinal Fractures | interventions — Kyphoplasty

STUDY DESIGN:
Intervention Model Description: Prospective Rondomized Open Blinded End Point
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kyphoplasty with Titanium spheres (Experimental): Patients treated with kyphoplasty with baloons and insertion of titanium microspheres inside the body vertebra.
  Interventions: Device: Kyphoplasty with insertion of Sctructured Titanium Microspheres
- Kyphoplasty with Polymethylmethacrilate (Active Comparator): Patients treated with Kyphoplasty with baloons and insertion of Polymethylmetacrylate inside the body vertebra.
  Interventions: Device: Kyphoplasty with Polimethylmetacrilate (convetional surgery)

INTERVENTIONS:
Device: Kyphoplasty with insertion of Sctructured Titanium Microspheres — Under fluoroscophy, we introduce a transpeduncolar trocar inside the vertebral body where is performed a kyphoplasty with insertion of baloons. When the dome is cretated we introduce structured titanium microspheres until the dome is full of material.
  Arms: Kyphoplasty with Titanium spheres
Device: Kyphoplasty with Polimethylmetacrilate (convetional surgery) — Under fluoroscophy, we introduce a transpeduncolar trocar inside the vertebral body where is performed a kyphoplasty with insertion of baloons. When the dome is cretated we introduce Polimethylmetacrilate until the dome is full of material.
  Arms: Kyphoplasty with Polymethylmethacrilate

SUMMARY:
The aim of the trial is to study efficacy and safety of Kyphoplasty technique with porous titanium microspheres in patients with type A vertebral body fracture (according to Magerl classification).

DETAILED DESCRIPTION:
Randomized controlled open trial with P.R.O.B.E. design (Prospective Randomized Open, Blinded End-point)

Objective:

The aim of the trial is to study efficacy and safety of Kyphoplasty technique with porous titanium microspheres in patients with type A vertebral body fracture (according to Magerl classification).

All consecutive eligible patients, belonging to the Neurosurgery Unit of A.R.N.A.S. Civico Hospital, in Palermo, will be included in the pilot study: 10 patients will be recruited for the treatment arm and 10 patients for the control arm.

* Patients aged between 18 and 80 years.
* Diagnosis of vertebral body fracture, type A (according to Magerl classification) in particular A.1, A.2 and A.3.1.
* Absence of ligamentous structures lesion and / or invasion of the spinal canal, confirmed by RX TC and NMR.
* Refusal to sign informed consent,
* Diagnosis different from those established by inclusion criteria.
* Age under 18 years.
* Age over 80 years.
* Presence of ligamentous structures lesion and / or invasion of the spinal canal confirmed by RX, TC and NMR.

For each patient will be evaluated:

* Spine RX
* CT of the spinal layer (or Spine CT)
* Spine MRI
* Roland Morris Disability (for the assessment of low back pain)
* EQ-5D (health questionnaire)
* Denis Work Scale (for the assessment of working conditions)
* VAS (for pain assessment)
* The statistical analysis will be performed using the SPSS software vers. 12.0 (SPSS Inc., Chicago, IL, United States). The study data will be collected pursuant to and for the purposes of articles 13 and 23 of the D. L.gs. n. 196/2003.

The study will be performed according to the rules established by the principles of Good Clinical Practice (as per Ministerial Decree of 07/15/97) and according to the principles gathered in the Helsinki Declaration (52 nd WMA General Assembly version, Edimburgh, Scotland, October 2000 ).

The clinical practices are performed according to the most recent recommendations of the World Medical Assembly (Declaration of Helsinki, 1964, and subsequent amendments).

ELIGIBILITY:
Inclusion Criteria:

* Magerl Type A Thoracolumbar fracture with no neurological deficits
* Age>18yy and < 80yy
* No ligament lesions

Exclusion Criteria:

* age < 18yy or > 80yy
* Ligament lesions
* refusal to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-09-25 (Estimated); Study Completion 2020-10-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of prototype device usage, as assessed by Change from baseline in post-surgical complication rate at 1 month. | 1 month post operative control
  Demonstrate if the prototype device is useful.

SECONDARY OUTCOMES:
Visual analogical Scale (VAS) and changing in time. | immediate, follow-up at 1-3-6 months after trauma
  Visual analogical Scale (VAS) from 0 to 10. Decreasing of VAS, compared to base line, will be considered a good point.
Pre, Post operation Vertebra height and changing in time | immediate, follow-up at 1-3-6 months after trauma
  Comparing Vertebra height in cm before and after surgery. Good height restoration will be considered a good point.
Acquired kyphosis | 6 months after trauma
  Cobb angle measurement. No angle acquisition it will be considered as a good point.
Ostheogenesis | 6 months after trauma
  Induced osteogenesis investigated by Bone Scintigraphy. Osteoinduction will be considered as positive point.

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Costantino, Palermo, PA, Italy

IPD SHARING:
Plan to Share IPD: Undecided